CLINICAL TRIAL: NCT05857176
Title: Assessment of Safety and Satisfaction Toward COVID-19 Vaccines: A Cross-sectional Study.
Brief Title: Assessment of Safety and Satisfaction Toward COVID-19 Vaccines.
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Other Study IDs: COVID-19 vaccines Perception
Record Dates: First submitted 2023-05-10; First posted 2023-05-12 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Vaccine Adverse Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID-19 Vaccine questionnaire — An online questionnaire, designed on Google Forms, was written in Arabic language and delivered to participants via social media (primarily Facebook, WhatsApp and Linkedin).
  Other Names: Google form questionnaire

SUMMARY:
This is a cross-sectional, web-based online survey done with the use of a Google Form-questionnaire to gather information from the general public regarding their knowledge, satisfaction, and tolerability about the COVID-19 vaccine.

DETAILED DESCRIPTION:
* A cross-sectional study was conducted. The subjects participating in the study are residents in Egypt.
* An online questionnaire, designed on Google Forms, was written in Arabic language and delivered to participants via social media (primarily Facebook, WhatsApp and Linkedin).
* The questionnaire comprised two categories of inquiries. The first is demographic data of the subject. The second is questions about COVID-19 vaccine-related data, such as whether had taken the vaccine or not, the type of vaccine administered, side effects encountered from the vaccine , if got enough information regarding the vaccine and where obtain the vaccine information from and if reluctant to taking the vaccine and the reasons for hesitancy. All participants were permitted to terminate the survey at any time of the study.

ELIGIBILITY:
Inclusion Criteria:

* all adults (age ≥ 18 years) complete the questionnaire were considered eligible to participate in the survey.

Exclusion Criteria:

* Incomplete questionnaires were excluded from the final analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects participating in the study are residents in Egypt who complete the online questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
headache incidence | 3 month
  Pecentage
fever incidence | 3 month
  Pecentage
fatigue incidence | 3 month
  Pecentage
pain at site of injection incidence | 3 month
  Pecentage

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass. Prof., Principal Investigator — Damanhour University
Locations (1):
- Rehab Hussein Werida, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malik A, Malik J, Ishaq U. Acceptance of COVID-19 vaccine in Pakistan among health care workers. PLoS One. 2021 Sep 15;16(9):e0257237. doi: 10.1371/journal.pone.0257237. eCollection 2021. PMID 34525110
- [Background] Lazarus JV, Ratzan SC, Palayew A, Gostin LO, Larson HJ, Rabin K, Kimball S, El-Mohandes A. A global survey of potential acceptance of a COVID-19 vaccine. Nat Med. 2021 Feb;27(2):225-228. doi: 10.1038/s41591-020-1124-9. Epub 2020 Oct 20. PMID 33082575